CLINICAL TRIAL: NCT02611921
Title: Intranasal Ketamine Use in Autism Spectrum Disorder: A Placebo-Controlled Crossover Pilot Study
Brief Title: Study of Intranasal Ketamine for Social Impairment in Autism Spectrum Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Roivant Sciences, Inc. (Industry); Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-2494
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Ketamine; Social Impairment; Autism; Autistic Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crossover Group: Ketamine verses Placebo (Experimental): Phase 1: Two ascending doses of intranasal ketamine
  Two week washout
  Phase 2: Two doses of placebo
  Interventions: Drug: Ketamine; Drug: Placebo
- Crossover Group: Placebo verses Ketamine (Experimental): Phase 1: Two doses of placebo
  Two week washout
  Phase 2: Two ascending doses of intranasal ketamine
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine will be compounded into a mucosal atomization device and self-administered or administered with assistance of a caregiver/study coordinator
  Other Names: Ketalar
Drug: Placebo — Placebo will delivered as an atomized saline spray which will be self-administered or administered with assistance of a caregiver/study coordinator
  Other Names: Saline

SUMMARY:
The purpose of the study is to determine if intranasal ketamine shows initial evidence of safety, tolerability and efficacy for the treatment of social impairment in individuals with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
To address the significant need for effective treatment of core symptoms of Autism Spectrum Disorder (ASD), this trial is designed as a double-blind, placebo-controlled crossover pilot study of intranasal ketamine in 24 individuals with ASD ages 12- 30 years using a novel quantitative eye-tracking outcome measure to assess impact of the drug on social impairment. Additionally, to develop a ketamine-focused personalized medicine approach in ASD, the investigators will include pharmacokinetic, molecular pharmacodynamic, and electrophysiological assessments into initial systematic study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 30 years old.
* Weight equal to or greater than 50 kg.
* General good health as determined by physical exam, medical history, laboratory work up, and EKG.
* Diagnostic and Statistical Manual of Mental Disorders 5th Edition diagnosis of autism spectrum disorder (not associated with Fragile X Syndrome or other known genetic syndrome) as confirmed by the Autism Diagnostic Observation Schedule at screen or previous (within last 5 years) if available.
* Valid Intelligence Quotient (IQ) score greater than or equal to 50 as confirmed via testing (Leiter-3) at screen or previous (within last 5 years, any valid testing acceptable).
* Clinical Global Impressions-Severity score of 4 (Moderately Ill).
* Score of 10 on the Social Withdrawal subscale of the Aberrant Behavior Checklist.
* Stable dosing of all concomitant psychotropic medications for five half-lives prior to screening visit and during the study.
* Presence of parent/guardian or significant other or caregiver willing to serve as informant for behavioral outcome measures.

Exclusion Criteria:

* Presence of co-morbid schizophrenia, schizoaffective disorder, bipolar disorder with psychosis, bipolar disorder or psychosis not otherwise specified. Comorbid diagnoses determined by psychiatrist clinical interview and use of Diagnostic and Statistical Manual of Mental Disorders 5th Edition diagnostic criteria.
* History of drug or alcohol abuse.
* Presence of cardiac disease including coronary artery disease, congestive heart failure, or uncontrolled hypertension per medical history (individuals with ≥ 2 blood pressure readings of ≥140/90 during screen/baseline will be excluded).
* Airway instability, tracheal surgery, or tracheal stenosis per medical history.
* Central nervous system masses or hydrocephalus per medical history.
* Porphyria, thyroid disorder, or thyroid medication use per medical history.
* Glaucoma or other cause of increased intraocular pressure per medical history.
* Allergy to ketamine.
* Current use of drugs with concomitant modification of non-competitive N-methyl-D-aspartate glutamate activity (acamprosate, amantadine, memantine, d-cycloserine etc.)
* For female subjects of child bearing potential, a positive pregnancy test.
* Any major chronic medical or chronic respiratory illness considered to be uncontrolled by the Principal Investigator.
* Inability to tolerate study procedures or study drug per the discretion of the Principal Investigator.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Change in Social Withdrawal subscale score of the Aberrant Behavior Checklist (ABC) | Social withdrawal subscale change from baseline to final visit on day 35 ± 2 days
  The ABC is the gold standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials.

SECONDARY OUTCOMES:
Change in the Clinician-rated CGI Improvement scale (CGI-I) | CGI-I change from baseline to final visit on day 35 ± 2 days
  The CGI-I is a 7-point scale designed to measure symptomatic change at a specific time as compared to baseline. The CGI-I will be focused on the target symptoms of social impairment. CGI-I is a gold standard measure of potential change with treatment in placebo- controlled pharmacotherapy trials in ASD

CONTACTS AND LOCATIONS:
Overall Officials: Logan K Wink, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No